CLINICAL TRIAL: NCT00109993
Title: Phase II Clinical Trial Incorporating Alemtuzumab (Campath-1H) in Combination With FK506 and Methylprednisolone for Treatment of Severe Acute Graft vs Host Disease
Brief Title: Campath-1H + FK506 and Methylprednisolone for GVHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mary Laughlin, MD, Ireland Cancer Center at University Hospitals Case Medical Center,Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE1Z04; P30CA043703 (NIH); CASE-CWRU-1Z04 (Other: Case Comprehensive Cancer Center); CWRU-060419; CASE-1Z04 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; refractory multiple myeloma; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage II ovarian epithelial cancer; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, T-Cell, Cutaneous; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Leukemia, Hairy Cell | interventions — Alemtuzumab; Methylprednisolone; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: alemtuzumab — alemtuzumab IV over 2 hours on days 4-6, 18, and 32
Drug: methylprednisolone — methylprednisolone IV on days 1-3 and then orally or IV on days 4-14
Drug: tacrolimus — tacrolimus IV continuously on days 1-7 and then orally once or twice daily on days 8-180, followed by a taper in the absence of chronic graft-vs-host disease

SUMMARY:
RATIONALE: Alemtuzumab, tacrolimus, and methylprednisolone may be an effective treatment for graft-versus-host disease caused by a donor stem cell transplant.

PURPOSE: This phase II trial is studying how well giving alemtuzumab together with tacrolimus and methylprednisolone works in treating acute graft-versus-host disease in patients who have undergone donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 4-week rate of complete response in patients with severe acute graft-vs-host disease (GVHD) treated with alemtuzumab, tacrolimus, and methylprednisolone within 100 days after undergoing allogeneic stem cell transplantation.

Secondary

* Determine the best response at 4 and 12 weeks in patients treated with this regimen.
* Determine 6-month survival of patients treated with this regimen.
* Determine the rate of infectious complications in patients treated with this regimen.
* Determine rate of chronic GVHD in patients treated with this regimen.

OUTLINE: This is an open-label, single-blind, multicenter study.

Patients receive methylprednisolone IV on days 1-3 and then orally or IV on days 4-14; tacrolimus IV continuously on days 1-7 and then orally once or twice daily on days 8-180, followed by a taper in the absence of chronic graft-vs-host disease; and alemtuzumab IV over 2 hours on days 4-6, 18, and 32. Treatment continues in the absence of unacceptable toxicity or the development of serious infection.

After completion of study treatment, patients are followed at 2 and 4 weeks.

PROJECTED ACCRUAL: A total of 9-34 patients will be accrued for this study within 8-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute graft-vs-host disease (GVHD)

  * Clinical grade C or D disease

    * No grade C disease with single organ skin involvement
* Has undergone allogeneic stem cell transplantation within the past 100 days

  * Absolute neutrophil count > 500/mm^3 (donor-derived [> 60% by peripheral blood lymphocyte chimerism analyses])
* No development of GVHD after prior donor lymphocyte infusion
* Must have received prior prophylactic cyclosporine or tacrolimus at the onset of acute GVHD

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* No serologic evidence of active hepatitis B or C infection

Renal

* Creatinine ≤ 3.5 mg/dL
* No requirement for dialysis

Cardiovascular

* No requirement for vasopressors

Pulmonary

* No requirement for a ventilator

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No known HIV positivity
* No active uncontrolled infection
* No other organ dysfunction

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Graft-vs-host disease response | 1, 2, 3, and 4 months

SECONDARY OUTCOMES:
Incidence of serious infections by clinical, radiologic, and microbiologic assessments | 1,2,3, and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Laughlin, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (6):
- United States (6):
  - Mt. Sinai Medical Center, New York, New York
  - Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Texas Transplant Institute, San Antonio, Texas